CLINICAL TRIAL: NCT01659970
Title: A Prospective Cohort Study Assessing the Efficacy and Safety of Tarceva in 2nd Line in Patients With Locally Advanced or Metastatic Squamous Non-small Cell Lung Cancer (NSCLC)
Brief Title: PEPITA Study: An Observational Study of Tarceva (Erlotinib) in Second Line in Patients With Locally Advanced or Metastatic Squamous Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28195
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the efficacy and safety of Tarceva (erlotinib) in second line in patients with locally advanced or metastatic squamous non-small cell lung cancer (NSCLC) after failure of first line platinum-based chemotherapy. Eligible patients will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically confirmed advanced (Stage IIIB) or metastatic (Stage IV) squamous non-small cell lung cancer after failure of first-line platinum-based chemotherapy
* Patients for whom the treating physician has decided to initiate treatment with Tarceva

Exclusion Criteria:

* Mixed non-small cell and small-cell lung carcinoma or mixed squamous cell carcinoma with predominant adenocarcinoma component
* Current participation in a clinical trial evaluating an anticancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic squamous NSCLC initiating 2nd line treatment with Tarceva
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 years

SECONDARY OUTCOMES:
Clinical/demographic patients characteristics at baseline | 2 years
Treatment schedules: Dose/duration/modifications/interruptions | 2 years
Overall survival | 2 years
Safety: Incidence of adverse events | 2 years
Quality of life: FACT-L version 4 questionnaire | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (93):
- France (93):
  - Abbeville
  - Agen
  - Aix-en-Provence
  - Amiens
  - Angers
  - Antibes
  - Armentières
  - Aulnay-sous-Bois
  - Bar-le-Duc
  - Bayonne
  - Beuvry
  - Bordeaux
  - Boulogne-Billancourt
  - Bourg-en-Bresse
  - Brive-la-Gaillarde
  - Bron
  - Bry-sur-Marne
  - Carcassonne
  - Castres
  - Chalon-sur-Saône
  - Chambéry
  - Charleville-Mézières
  - Chaumont
  - Chauny
  - Clamart
  - Clermont-Ferrand
  - Colmar
  - Compiègne
  - Créteil
  - Dijon
  - Draguignan
  - Dunkirk
  - Ermont
  - Épernay
  - Férolles-Attilly
  - Forbach
  - Gap
  - Gleizé
  - Gonesse
  - La Rochelle
  - La Source
  - La Tronche
  - Lagny-sur-Marne
  - Le Mans
  - Le Puy-en-Velay
  - Lille
  - Limoges
  - Lisieux
  - Longjumeau
  - Lorient
  - Lyon
  - Manosque
  - Mantes-la-Jolie
  - Mareuil-lès-Meaux
  - Marseille
  - Meaux
  - Metz
  - Metz-Tessy
  - Mont-de-Marsan
  - Montpellier
  - Nancy
  - Nantes
  - Narbonne
  - Neuilly-sur-Seine
  - Paris
  - Perpignan
  - Pierre-Bénite
  - Poitiers
  - Pontoise
  - Quimper
  - Rambouillet
  - Reims
  - Rennes
  - Rouen
  - Saint-Dié
  - Saint-Dizier
  - Saint-Jean
  - Saint-Laurent-du-Var
  - Saint-Omer
  - Saint-Priest-en-Jarez
  - Saint-Quentin
  - Saintes
  - Strasbourg
  - Thionville
  - Thonon-les-Bains
  - Toulon
  - Toulouse
  - Tours
  - Valence
  - Vandœuvre-lès-Nancy
  - Vannes
  - Verdun
  - Vénissieux